CLINICAL TRIAL: NCT06270797
Title: Pre-anesthesia Imaging-based Respiratory Assessment and Analysis
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20230184
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2023-12

CONDITIONS: Clinical Decision Support System
Keywords: knowledge graph; artificial intelligence; Enhanced Recovery After Surgery
MeSH Terms: interventions — Intubation; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal intubation: during general anesthesia, normal intubation without any difficult airway or difficult intubation were recorded in the note.
  Interventions: Procedure: intubation for general anesthesia
- difficult airway or difficult intubation: during general anesthesia, any type of difficult airway or difficult intubation were recorded in the note.
  Interventions: Procedure: intubation for general anesthesia

INTERVENTIONS:
Procedure: intubation for general anesthesia — routine intubation for general anesthesia

SUMMARY:
This study is to establish a preoperative respiratory imaging assessment database and develop a difficult intubation risk prediction model and further risk analysis. We attempt to construct it into a pre-anesthesia intubation risk assessment software as the clinical decision support system.

DETAILED DESCRIPTION:
Anesthesia respiratory assessment is an important issue for anesthesiologists to evaluate the respiratory status and airway management of patients before surgery. The American Society of Anesthesiologists (ASA) updated its guidelines in 2022, emphasizing the importance of comprehensive respiratory assessment in the guidelines.

Various risk factors have been proposed in past literature for discussion, and corresponding to these risk factors, there is currently no single factor that can predict difficult intubation completely. Existing investigations into difficult intubation factors mostly focus on high-risk populations, including patients with morbid obesity, where significant differences have been identified but not developed into predictive models.

With the rapid development of AI-related technologies in recent years, numerous image-related AI frameworks have been proposed. In recent years, attempts have been made to combine various clinical risk factors using machine learning methods to create automated prediction models for difficult intubation. However, their effectiveness has not met expectations, reflecting the significant clinical problem of difficulty in prediction that remains unresolved.

This study is an observational study aimed at analyzing and establishing patient image data, refining various data engineering techniques, and optimizing existing prediction model frameworks to enhance their medical value. Additionally, the focus of this project will be on establishing more prediction models to improve existing clinical decision support systems.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing general anesthesia
* Patients who can undergo pre-anesthetic consultation and airway examination.

Exclusion Criteria:

* Patients unable to undergo pre-anesthetic consultation and airway examination.
* Patients requiring emergency surgery.
* Vulnerable populations.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing regular general anesthesia with pre-anesthetic consultation and airway examination.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
A pre-anesthesia evaluation | pre-anesthetic consultation about 20 min
  The examination includes airway assessment and dental evaluation.
Perform non-invasive imaging capture. | pre-anesthetic consultation about 5 min
  The capture involves non-invasive imaging of the patient's facial features through standard basic photography, excluding any additional radiographic imaging examinations.The patient's images will be stored in de-identified form.
difficult intubation prediction | after pre-anesthetic consultation about 5 min
  The prediction of difficult intubation from pre-anesthesia evaluation and non-invasive imaging capture

SECONDARY OUTCOMES:
time to successfully extubate the nasotracheal tube after anesthesia | from the end of surgery to the post-anesthesia care, assessed up to one hour
  early extubation allowable
safely discharged from post-anesthesia care unit (postoperative recovery room) | 2 hours
  as calculating the time from patient is delivered to postoperative recovery room to be safely discharged from recovery room by using the aldrete scores (activities level, respiration, circulation, conscious level, oxygenation) full back to pre-operative level or ten scores.
side effects and adverse events | intraoperative and postoperative stages, assessed up to 48 hours
  records any abnormal surgical or anesthesia related findings during this admission

CONTACTS AND LOCATIONS:
Overall Officials: Kuang-I Cheng, MD,Phd, Study Director — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided